CLINICAL TRIAL: NCT01112345
Title: A Multicentre, Non Interventional, Non Randomized, Observational Study for the Assessment of Compliance and Persistence With Rebif® Therapy of Patients With Relapsing-Remitting Multiple Sclerosis as Well as for the Evaluation of Potential Factors Influencing These Parameters, in Real Life Clinical Practice
Brief Title: An Observational Study for the Assessment of Compliance and Persistence to Rebif® Therapy of Patients With Relapsing-remitting Multiple Sclerosis (MS) and Evaluation of Potential Factors Influencing These Parameters
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck A.E., Greece (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 701068-513
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Interferon-beta
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The present study aims to assess the adherence to therapy with interferon beta-1a (Rebif®) and at investigating potential factors that are involved in its outcome, in a representative sample of patients with relapsing remitting multiple sclerosis (RRMS), under real life conditions.

DETAILED DESCRIPTION:
In the relapsing-remitting type of the disease the objective of the therapy is the reduction of relapse rate, duration and severity, as well as the delay of transition to the progressive form of the disease. Subjects' adherence to long-term therapy of MS plays a pivotal role in the optimization of therapeutic outcome and maximization of the derived clinical benefit for the treated subjects. Rebif current formulation has been developed by assessing and refining the physicochemical characteristics of existing formulations aiming at further improving product's tolerability profile. Studies performed for the assessment of Rebif have demonstrated a 3-fold reduction in injection site reactions as well as improved overall tolerability and safety profile.

This is a multicentre, prospective, non interventional, non randomized, open label study for the assessment of the adherence to therapy with Rebif of subjects with RRMS. The participating subjects shall be already on treatment with (Rebif) prior to their enrolment into the study, according to the approved Summary of Product Characteristics (SPC) and the clinical, imaging and laboratory findings of the disease, as evaluated by their treating physician, in real life clinical practice. Data will be collected retrospectively from a sample of 150 subjects' medical files and through questions that will be posed to the subjects, and prospectively during the course of the study. The total duration of the study is estimated to be 18 months.

OBJECTIVES

Primary objective:

* To assess the compliance and persistence with Rebif therapy in MS subjects, after six months of therapy, in "real life" clinical settings in Greece

Secondary objective:

* To investigate the potential factors influencing compliance and persistence to Rebif therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented diagnosis of RRMS according to the Mc Donald criteria (2005)
* Subjects who have already been administered therapy with IFN b-1a (Rebif) according to the approved product's Summary of Product Characteristics (SPC), at least two weeks and not longer than six weeks prior to their enrolment into the study
* Subjects of both genders, aged between 18 - 65 years (inclusive)
* Expanded Disability Status Scale (EDSS) score < 6 (inclusive) at baseline (before Rebif therapy initiation)
* Subjects who are able to read and understand the Patient Information Leaflet
* Subjects who have signed the Informed Consent Form
* Subjects who are willing and capable to comply will all study requirements and procedures.

Exclusion Criteria:

* Subjects that meet any of the contraindications to the administration of the study drug according to the approved SPC
* Subjects with primary progressive or secondary progressive form of MS
* Subjects who have been treated with Rebif for less than two weeks and more than six weeks before their enrollment into the study
* Subjects who had been receiving any therapy for MS (other disease modifying drugs, immunomodulatory and/or immunosuppressive agents) within three months before Rebif therapy commencement
* History of any chronic pain syndrome
* Current or past (during the preceding two years) history of alcohol or drug abuse
* Women who are pregnant or breastfeeding or of childbearing potential that do not use any medically accepted method of contraception
* Subjects who are currently participating or had participated in another clinical trial during the last three months prior to their enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with documented diagnosis of RRMS according to the McDonald criteria (2005)
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Assessment of subjects' compliance with physicians' instructions on the proper use of the treatment | Preceding 2 weeks prior to subjects enrolment into the study
  Evaluation of the actual number of injections administered during the preceding 2 weeks prior to subjects' enrolment into the study
Assessment of subjects' compliance with physicians' instructions on the proper use of the treatment after 6 months of therapy | From preceding 2 weeks prior to the first visit (Month 1) till the final visit (Month 6) of the study
  Evaluation of the number of injections actually administered over the preceding 2 weeks prior to the first and the final visit of the study
Assessment of subjects' persistence to therapy | Since subjects' enrolment until final study visit (Month 6)
  Assessment will include recording of the number of days under treatment since subjects' enrolment into the study and until the performance of the study final visit, at Month 6.

SECONDARY OUTCOMES:
Assessment of the factors and their potential correlation with the defined subjects' compliance and persistence to therapy | Subjects' enrollment to final study visit (Month 6)
  Subject's training regarding proper administration of the study drug and proper use of auto-injector of the study drug (Rebiject II); implementation by subject of the recommendations for treatment administration and instructions on the proper use of device (via prefilled syringe or auto-injector); prophylactic use of non steroidal anti-inflammatory drugs (NSAIDs); reasons for missed injections; EDSS score at baseline; relapse history prior to Rebif therapy initiation; MS treatments received by the subject during the preceding year before Rebif therapy commencement

CONTACTS AND LOCATIONS:
Overall Officials: Michalis Arvanitis, MD, Study Director — Merck A.E., Greece
Locations (1):
- Henry Dunant Hospital - IRB, Athens, Greece

REFERENCES:
- [Background] Manfredonia F, Pasquali L, Dardano A, Iudice A, Murri L, Monzani F. Review of the clinical evidence for interferon beta 1a (Rebif) in the treatment of multiple sclerosis. Neuropsychiatr Dis Treat. 2008 Apr;4(2):321-36. doi: 10.2147/ndt.s476. PMID 18728744
- [Background] Murdoch D, Lyseng-Williamson KA. Subcutaneous recombinant interferon-beta-1a (Rebif): a review of its use in relapsing-remitting multiple sclerosis. Drugs. 2005;65(9):1295-312. doi: 10.2165/00003495-200565090-00010. PMID 15916455
- [Background] Gold R, Rieckmann P, Chang P, Abdalla J; PRISMS Study Group. The long-term safety and tolerability of high-dose interferon beta-1a in relapsing-remitting multiple sclerosis: 4-year data from the PRISMS study. Eur J Neurol. 2005 Aug;12(8):649-56. doi: 10.1111/j.1468-1331.2005.01083.x. PMID 16053475
- [Background] Cramer JA, Cuffel BJ, Divan V, Al-Sabbagh A, Glassman M. Patient satisfaction with an injection device for multiple sclerosis treatment. Acta Neurol Scand. 2006 Mar;113(3):156-62. doi: 10.1111/j.1600-0404.2005.00568.x. PMID 16441244